CLINICAL TRIAL: NCT02138461
Title: Subjective Patient Assessment Comparing Overall Tolerability and Satisfaction of a Prostaglandin Analogue Including Either Bimatoprost 0.01% or Latanoprost.
Brief Title: Tolerability of Bimatoprost 0.01% vs Latanoprost Eye Drops
Status: Completed | Type: Observational
Sponsor: MDbackline, LLC (Other)
Collaborators: Allergan (Industry)
Responsible Party: Sponsor
Other Study IDs: JH-ALG-MDB-1301
Record Dates: First submitted 2014-05-09; First posted 2014-05-14 (Estimated); Results first posted 2014-09-25 (Estimated); Last update posted 2014-09-25 (Estimated); Status verified 2014-09

CONDITIONS: Glaucoma
Keywords: glaucoma; bimatoprost; latanoprost; tolerability
MeSH Terms: conditions — Glaucoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: None Retained — Note patients will be recruited to fill out a questionnaire, describing their symptoms related to glaucoma use drops. In this study, we are examining only patients taking either bimatoprost or latanoprost, thus 2 cohorts. However, this is not an interventional study, and there will be only one study visit (enrollment and questionnaire at the same time) and no change in the patient's prescribed therapy.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- bimatoprost: These patients take bimatoprost topically for glaucoma.
- latanoprost group: These patients take latanoprost topically for glaucoma.

SUMMARY:
This study examines patient perceptions regarding the tolerability of two classes of glaucoma medication: bimatoprost and latanoprost.

DETAILED DESCRIPTION:
Patients enrolled in this study completed a validated survey instrument (COMTOL) examining tolerability of topically applied ophthalmic medications that they are already taking in their regular course of care for glaucoma. The purpose of the study is to determine whether side effects and symptoms of the drugs already being taken cause problems with activities of daily living.

ELIGIBILITY:
Inclusion Criteria:

* Patients with glaucoma taking either bimatoprost or latanoprost

Exclusion Criteria:

* patients taking other medication or with other causes for ocular surface symptoms

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients taking either study medication for glaucoma.
Sampling Method: Probability Sample
Enrollment: 211 (Actual)
Dates: Start 2013-10; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John A. Hovanesian, MD, Principal Investigator — UCLA Jules Stein Eye Institute; Savak Teymoorian, MD, Principal Investigator — Harvard Eye Associates
Locations (1):
- Harvard Eye Associates, Laguna Hills, California, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Bimatoprost | Latanoprost Group
Started | 101 | 110
Completed | 101 | 110
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Bimatoprost | Latanoprost Group | Total
Number analyzed (Participants) | 101 | 110 | 211
Age, Continuous [Mean (Standard Deviation); unit: years] | 75.3 (12.0) | 73.4 (12.1) | 74.4 (12.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 63 | 56 | 119
  Male | 38 | 54 | 92
Region of Enrollment [Number; unit: participants]
  United States | 101 | 110 | 211

OUTCOME MEASURES:

1. Primary Outcome: Tolerability of Medications as Measured by the COMTOL Validated Instrument
Description: Patients who are already taking the medications of interest will be enrolled from a general ophthalmology practice. Immediately after consenting to participate, they will complete a validated survey instrument called the Comparison of Ophthalmic Medication for Primary Outcome Measure Tolerability (COMTOL) questionnaire (Ophthalmology 1997; : 104:334-342). Because this study will not be a crossover trial design, and patients will only continue taking the medications they were prescribed in the course of their glaucoma therapy, the modified version will eliminate questions in the COMTOL related to subjective comparison of two medications and instead focus on tolerability of the single medication being taken by test subjects.
Time Frame: at the time of enrollment in the clinic, patients will immediately complete the questionnaire and exit the study
Measure: Number; unit: percentage of patients
Arm/Group | Bimatoprost | Latanoprost Group
Number analyzed (Participants) | 101 | 110
percentage of patients
  Bothered by Itching More than "A Little" | 23 | 50
  Bothered by Burning/Stinging More Than "A Little" | 26 | 29
  Bothered by Redness More Than "A Little" | 31 | 42
  Bothered by Dry Eyes More Than "A Little" | 47 | 54

ADVERSE EVENTS:
Arm/Group | Bimatoprost | Latanoprost Group
Serious Adverse Events (participants affected / at risk) | 0/101 | 0/110
Other Adverse Events (participants affected / at risk) | 0/101 | 0/110

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No